CLINICAL TRIAL: NCT05611580
Title: Reducing Chronic Disease Risk Among Rural Adults
Brief Title: Rural Chronic Disease Risk Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Laurie Abbott, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003258
Record Dates: First submitted 2022-10-31; First posted 2022-11-10 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Chronic Disease; Risk Reduction
Keywords: chronic disease; health promotion; risk reduction
MeSH Terms: conditions — Chronic Disease; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The participant in the control group receive usual care.
- Intervention (Experimental): The participants in the intervention group received the chronic disease risk reduction intervention.
  Interventions: Behavioral: Chronic Disease Risk Reduction

INTERVENTIONS:
Behavioral: Chronic Disease Risk Reduction — The intervention involves education information about chronic diseases and way to reduce risk for developing chronic diseases and/or decrease worsening of existing conditions.
  Arms: Intervention

SUMMARY:
This study tests a web-based chronic disease risk reduction lifestyle medicine intervention among rural adults.

DETAILED DESCRIPTION:
The impact of chronic diseases has important implications for public health presently and in the future. The prevalence of chronic diseases is expected to rise with subsequent increases in mortality, morbidity, and health care costs. This proposed pilot project involves testing an adapted evidence-based lifestyle medicine (health promotion and disease risk reduction) curriculum using a web-based delivery format and determine its impact and efficacy among rural participants. The project is expected to contribute to improved human health by promoting healthy behaviors that reduce the development, progression, and exacerbation of chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years of age,
2. reside in a rural southern county (RUCC 4-9),
3. speak, write, and understand English,
4. have access to a computer with internet service or smartphone with cellular data,
5. have the ability to access the Zoom platform, and f) have at least one chronic disease risk factor or diagnosis (diabetes, prediabetes, overweight, smoker, hypertension, family history of cancer, diabetes, heart disease, elevated cholesterol level, overweight or obese, etc.).

Exclusion Criteria:

* not from a rural area
* younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Produce and Vegetable Consumption from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention.
  Theory of Planned Behavior 5-a-day Questionnaire: The 12-item scale for measuring produce consumption had adequate internal reliability for attitudes (Cronbach"s a = .79), norms (a = .77), self-efficacy (a = .81), and intentions (a = .74) when tested among a diverse population. The range of possible scores for each of the subscales for this instrument varied for attitudes (3 to 28), norms and self-efficacy (3 to 21), and intentions (1 to 14).
  Higher scores indicate greater compliance with dietary recommendations.

SECONDARY OUTCOMES:
Change in Sleep from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention.
  The Pittsburgh Sleep Quality Index (PSQI): Sleep habits, Perceptions of sleep quality, quantity, and difficulties falling and staying asleep. 9-item Likert scale had good internal reliability (α = .83).
  Higher scores indicate better sleep quality.
Change in Stress from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention.
  Perceived Stress Scale: A 10-item, 5-point Likert scale, that had excellent internal consistency (α = 0.84-0.86). The items include perceptions of stress.
  Higher scores indicate greater perceptions of stress.
Change in Social Support from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention.
  Interpersonal Support Evaluation List-12 (ISEL-12): Perceived belonging, tangible, and appraisal support. 12-item Likert scale had excellent reliability (α = .90).
  Higher scores indicate greater social support.
Change in Social Support to Eat Better and Move More from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention.
  Social Support to Eat Better and Move More: Support from friends; Overall (α = 0.96); Subscales [informational (α = 0.97), emotional (α = 0.96), and encouragement (α = 0.97)].
  Higher scores indicate greater social support to eat better and move more.
Change in Well-being from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention.
  Well-being Scale: Measures well-being (α = 0.92) overall, and five subscales (α = 0.79 - 0.85). Higher scores indicate greater perceptions of personal well-being.
Change in Dietary Fat Intake from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention.
  Theory of Planned Behavior Dietary Fat Measure: The 14-item instrument containing Likert-type subscales used to ascertain dietary fat attitudes (a = .95), norms (a = .92), self-efficacy (a = .86), and intentions (a = .94) was considered highly reliable. The range of potential scores included 2 items for attitudes (2 to 14), 4 items for norms (4 to 28), 5 items for self-efficacy (5 to 35), and 3 items for intentions (3 to 21).
  Higher scores indicate greater compliance with following dietary fat recommendations.
Change in Exercise from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention.
  Theory of Planned Behavior Exercise Questionnaire: 10-item scale used to measure exercise evidenced good reliability for attitude (α = .84), norms (α = .83), and self-efficacy. (α = .79). Higher scores indicate greater indications of exercise determinants.
Change in Health Habits and Knowledge from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention..
  Intervention-specific; Diet, exercise, confidence, smoking, alcohol; knowledge of CVD & risk factors. Both scales (Health Habits and Health Knowledge) range from 0-100.
  Higher scores indicate greater knowledge about health information and performance of those behaviors.
Change in Physical Activity from Baseline to Post-intervention and 4 weeks post-intervention | Baseline, Post-intervention (six weeks from baseline), 4 weeks post-intervention (10 weeks from baseline), and six months post-intervention.
  International Physical Activity Quesionnaire (IPAQ): Measures physical activities and exercise intensity and time levels, work-related physical activity, transportation-related, etc. (α = .80).
  Higher scores indicate greater levels of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University College of Nursing, Tallahassee, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT05611580/ICF_000.pdf